CLINICAL TRIAL: NCT04220918
Title: Taste of Medicines in Children: Genetic Variation and Medication Adherence
Brief Title: Taste of Medicines in Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Monell Chemical Senses Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-016182; R01DC011287 (NIH)
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Medication Adherence; Medication Reaction
Keywords: pediatrics; personalized medicine; GWAS; Taste; Side effects; clindamycin
MeSH Terms: conditions — Medication Adherence; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salivary DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some but not all children will refuse to take medicine because of its taste, which can lead to substantial worsening of disease, antibiotic resistance, increased health care costs, and even death. The investigators are systematically assessing individual variation in the taste of liquid clindamycin among genotyped pediatric patients prescribed clindamycin for standard of care treatment, to determine whether (1) genetic variation underlies differences in taste ratings of the antibiotic; (2) initial taste responses, genetics, or both predict likelihood of side effects and medication non-adherence.

DETAILED DESCRIPTION:
Taste plays an integral role in whether a child accepts a medicine. Some children will like the taste of a given medicine and complete the full course of treatment, whereas others will strongly reject its taste, suffer taste-modulated side effects, or both. This study will systematically measure initial palatability and reactions to the first dose of an antibiotic (clindamycin, liquid formulation) by pediatric patients who are receiving clindamycin as part of their standard of care treatment. Saliva will be collected from all patients for GWAS. Taste response, tolerance of the medication, adherence and clinical outcomes will be assessed. Subjects will be followed to determine if they complete the prescribed medication regimen (adherence) and/or experience side effects (tolerability). Because medication-specific side effects have patient-specific variability, the investigators will determine whether the child's initial taste responses, genes, or both predict subsequent side effects and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Children age 3 to 12
* Child being treated in Children's Hospital of Philadelphia
* Being prescribed clindamycin liquid
* Parental/guardian permission (informed consent) and if appropriate, child assent
* Parent age 18 or older, or a minor permitted by state law to consent for their own participation and for the participation of their child
* Parent must have primary responsibility for the patient including biologic parents and adoptive parents (if legally allowed to consent to research)
* Parent must be English speaking and able to understand study materials

Exclusion Criteria:

* Unwilling or unable to produce saliva sample

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who are prescribed clindamycin liquid at the Children's Hospital of Philadelphia (CHOP).
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Palatability of clindamycin liquid | Immediately after dosing
  Taste ratings by the child using a hedonic face scale (scale = 1-5; 1=dislike a lot, 2=dislike a little, 3=neither like nor dislike, 4=like a little, 5=like a lot)
Palatability of clindamycin liquid | 5 minutes after dosing
  Taste ratings by the child using a hedonic face scale (scale = 1-5; 1=dislike a lot, 2=dislike a little, 3=neither like nor dislike, 4=like a little, 5=like a lot)
Palatability of clindamycin liquid | 10 minutes after dosing
  Taste ratings by the child using a hedonic face scale (scale = 1-5; 1=dislike a lot, 2=dislike a little, 3=neither like nor dislike, 4=like a little, 5=like a lot)
Taste reactivity of clindamycin liquid | Immediately after dosing for a total of 10 minutes
  Digital recordings will be analyzed for child's facial and body movements by blinded and trained reviewers

SECONDARY OUTCOMES:
Medication tolerance and side effects with clindamycin use | 5-14 day treatment regimen given two-three times a day
  Medication tolerance and side effects to medication will be measured through direct observation, parent report, and medical records
Treatment adherence | 5-14 day treatment regimen given two-three times a day
  Adherence to treatment course will be measured by parental report aided by a medication diary
Clinical outcomes | within 1 week after completion of therapy
  Clinical outcome of infection (cured on clindamycin vs not cured on clindamycin) will be measured through medical record review and parental report during follow-up interview
Genome-wide association | 3 years
  salivary DNA

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth D Lowenthal, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia; Julie A Mennella, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No